CLINICAL TRIAL: NCT03039452
Title: Feasibility and Initial Effects of High Intensity Interval Training on Knee Osteoarthritis: an Exploratory Evaluation on Metabolomics
Brief Title: High Intensity Interval Training in Osteoarthritis, Effects on Metabolomics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-0829; 1P2CHD086851-01 (NIH)
Record Dates: First submitted 2017-01-18; First posted 2017-02-01 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High intensity interval training (Experimental)
  Interventions: Behavioral: High intensity interval training

INTERVENTIONS:
Behavioral: High intensity interval training — Each training session will consist of a 3-5 minute warm-up, followed by 10 repetitions of 1-minute bouts at individualized training intensity with 1-minute rest periods.
  Other Names: Stationary bike

SUMMARY:
Purpose: The purpose of this study will be to examine the feasibility and acceptability of a 6-week high intensity interval training (HIIT) program in patients with knee OA symptoms ranging from mild to severe. A secondary purpose will be to evaluated changes in whole body metabolism induced by 6-weeks of HIIT.

Participants: Fifteen patients (age 40-70 yrs; BMI 20-35 kg/m²) with symptomatic knee OA

Procedures (methods): All participants will be assigned to the single-arm of the study in which all participants will receive 6 weeks of HIIT, delivered twice per week. Outcomes will be assessed at baseline and 6 weeks. The primary outcome will evaluate tolerability, feasibility, acceptability, compliance, and adherence to the HIIT program. Secondary outcomes will include whole body metabolism markers, inflammation, and a set of physical function including knee osteoarthritis symptomatic burden and pain, cardiorespiratory fitness, isometric knee extensor and flexor strength (factors associated with physical function and symptomatic knee OA progression), and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Must exhibit symptomatic knee OA (WOMAC > 31), radiographic evidence of tibiofemoral OA (2-4 Kellgren-Lawrence scale)
* Age 40-70 years
* Body mass index 20-35 kg/m²
* Cleared by study physician from 12 lead EKG and medical history review

Exclusion Criteria:

* Individuals diagnosed with a cardiovascular condition restricting exercise Individuals currently meeting Department of Health and Human Services Guidelines for Physical Activity (meeting >150 minutes of exercise per week)
* Individuals currently doing HIIT
* Individuals currently participating in physical therapy for knee OA
* Individuals currently participating in another OA intervention study
* Received a corticosteroid or hyaluronic acid injection involved in the knee in the previous 3 weeks or scheduled for during the intervention
* Diagnosis of gout in the knee
* Diagnosis of Rheumatoid arthritis
* Diagnosis of Fibromyalgia
* Other systemic rheumatic disease
* Severe dementia or other memory loss
* Active diagnosis of psychosis or uncontrolled substance abuse disorder
* Hospitalization for a stroke, heart attack, or heart failure, or had surgery for blocked arteries in the past 6 months
* Diabetics (medications include exogenous insulin)
* Total joint replacement knee surgery, other knee surgery, meniscus tear, or ACL tear in the past 12 months
* On a waiting list for total joint replacement
* Severely impaired hearing or speech
* Pregnant or planning to become pregnant in the next 8 weeks
* Inability to speak English
* Serious or terminal illness as indicated by referral to hospice or palliative care
* Nursing home residence
* Inability to ride a stationary bike
* Any other health problems that would prohibit safe participation in the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Feasibility - proportion of potential participants screened for the study who are enrolled | baseline
Feasibility - retention: proportion of enrolled participants retained at 6-weeks post testing | 6 weeks

SECONDARY OUTCOMES:
Compliance: average number of training session completed per week | 6 weeks
Adherence: total number of training session completed per week | 6 weeks
Adherence: total number of training weeks completed | 6 weeks
Whole body metabolism measured by insulin | 6 weeks
Whole body metabolism measured by amino acids | 6 weeks
Whole body metabolism measured by free fatty acids | 6 weeks
Whole body metabolism measured by an oral glucose tolerance test | 6 weeks
Inflammation measured from interleukin-6 and tumor necrosis factor alpha | 6 weeks
Change in Pain score from baseline to 6 weeks | baseline, 6 weeks
  Determined from WOMAC pain subscale (range 0-20)
Change in symptomatic burden score from baseline to 6 weeks | baseline, 6 weeks
  Determined from the total WOMAC (range 0-96)
Cardiorespiratory Fitness from peak oxygen consumption test | 6 weeks
Knee Strength (extensors and flexors) from dynamometry | 6 weeks
Body Composition from dual energy x-ray absorptiometry | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Applied Physiology Laboratory, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Smith-Ryan AE, Blue MNM, Anderson KC, Hirsch KR, Allen KD, Huebner JL, Muehlbauer MJ, Ilkayeva OR, Kraus VB, Kraus WE, Golightly YM, Huffman KM. Metabolic and physiological effects of high intensity interval training in patients with knee osteoarthritis: A pilot and feasibility study. Osteoarthr Cartil Open. 2020 Jun 10;2(4):100083. doi: 10.1016/j.ocarto.2020.100083. eCollection 2020 Dec. PMID 36474875